CLINICAL TRIAL: NCT06233383
Title: Developing an Approach to Implementing Breast Cancer Screening Using Clinical Breast Exam in the Primary Health Centers of Soweto, South Africa
Brief Title: Developing Screening Clinical Breast Examination Implementation Strategies in South Africa
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: 2000036834
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adopters: Individuals responsible for deciding to institute screening CBE in Soweto's primary care clinics (e.g., policymakers, clinic administrators, nurse managers)
- Implementers: Individuals responsible for actually performing the screening CBE in Soweto's primary care clinics (e.g., nurses, doctors, fieldworkers, clerical workers)
- Recipients: Individuals eligible for a screening CBE (e.g., women over the age of 40 years from the community surrounding study clinics)

SUMMARY:
The goal of this observational study is to engage with multilevel stakeholders to collaboratively and to systematically develop a suite of strategies for implementing breast cancer screening using clinical breast examination (CBE) in the primary health centers within the catchment area of Chris Hani Baragwanath Academic Hospital (Bara Hospital), Johannesburg, South Africa.

The main questions it aims to answer are: What barriers and facilitators exist to conducting screening CBE in Soweto's primary care setting and what implementation strategies would support CBE in primary care clinics?

Participants will:

* Allow observation of study clinic workflows
* Participate in focus group discussions regarding screening CBE implementation

ELIGIBILITY:
In order to be eligible for inclusion in the focus group discussions held with screening CBE "adopters" and "implementers," an individual must meet all of the following criteria:

1. Be an employee or volunteer working at a participating PHC OR Be an employee or volunteer working at South Africa's National Department of Health OR Be an employee or volunteer working with a non-governmental organization that performs breast cancer related activities within the catchment area of a participating PHC
2. Be willing to commit to keeping the content of focus group discussions confidential

In order to be eligible for inclusion in the focus group discussions held with screening CBE "recipients," an individual must meet all of the following criteria:

1. Be female
2. Be between the ages of 40 and 65 years
3. Be living within the catchment area of a participating PHC
4. Be willing to commit to keeping the content of focus group discussions confidential

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Focus group participants will consist of three categories: screening CBE "adopter" (e.g., clinic administrators/managers, department of health officials, etc), "implementers" (e.g., nurses, physicians, community health workers), and "recipients" (e.g., women from the community eligible for CBE screening and community breast cancer survivors).
  All participants will be drawn from the four study clinics in Soweto, South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Implementation Strategies Suite | 2 years
  A collection of strategies for implementing routine screening clinical breast examination in Soweto's primary care clinics.

SECONDARY OUTCOMES:
Intervention Domain Characteristics | 2 years
  Characteristics of routine clinical breast examination itself that are potential barriers and facilitators to screening implementation
Inner Setting Domain Characteristics | 2 years
  Characteristics of the primary care clinics that are potential barriers and facilitators to screening implementation
Outer Setting Domain Characteristics | 2 years
  Characteristics of both the community surrounding the clinics and the district-wide health system that are potential barriers and facilitators to screening implementation
Individuals Domain Characteristics | 2 years
  Characteristics of individuals involved in screening that are potential barriers and facilitators to screening implementation
Implementation Domain Characteristics | 2 years
  Characteristics of activities and strategies used to implement screening that are potential barriers and facilitators to screening implementation
Change Matrices | 2 years
  Matrices for all individuals relevant to implementation that define performance objectives and corresponding performance determinants

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O'Neil, MD, MPH, Principal Investigator — Yale University
Locations (1):
- University of Witwatersrand, Faculty of Health Sciences, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No
In order to comply with local legal requirements, individual participant data will not be available to other researchers.